CLINICAL TRIAL: NCT01146704
Title: Gastrointestinal Hormonal Regulation of Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: F7219-R
Record Dates: First submitted 2010-04-02; First posted 2010-06-17 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Proteins; Carbohydrates; Diet, High-Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Diet (Active Comparator): Standard protein diet group as control based on 0.5 gram protein per pound of lean body mass with same calories: 15% protein and 55% carbohydrate.
  Interventions: Dietary Supplement: Protein powder supplement, standard dosage based on 0.5 gram protein per pound of subject's lean body mass
- High Protein Diet (Active Comparator): High protein diet group based on 1 gram of protein per pound of lean body mass: 30% protein and 40% carbohydrate.
  Interventions: Dietary Supplement: Protein powder supplement, High Level Protein, based on 1 gram of protein per pound of lean body mass: 25% protein and 45% carbohydrate

INTERVENTIONS:
Dietary Supplement: Protein powder supplement, standard dosage based on 0.5 gram protein per pound of subject's lean body mass — Standard protein diet as control, based on 0.5 gram protein per pound of lean body mass, isocaloric (same number of calories) and consisting of 15% protein and 55% carbohydrate.
  Other Names: Standard Protein Diet
  Arms: Standard Diet
Dietary Supplement: Protein powder supplement, High Level Protein, based on 1 gram of protein per pound of lean body mass: 25% protein and 45% carbohydrate — High level of protein diet, based on 1 gram of protein per pound of subject's lean body mass, isocaloric (same number of calories) and consisting of 30% protein and 40% carbohydrate.
  Other Names: High Protein Diet
  Arms: High Protein Diet

SUMMARY:
The objective of this study is to test and determine whether a high protein diet is efficacious, safe and beneficial to curtail food intake and body weight in obese adult human patients and to establish whether neurohormonal mechanisms of a high protein diet induce an early signal of fullness or satiety in a relevant experimental model, focusing on activation of gastric vagal afferents.

DETAILED DESCRIPTION:
Obesity is a major cause of morbidity and mortality within the VA medical system accounting for the majority of cases of diabetes mellitus, hypertension, coronary artery disease and cerebrovascular accidents. An improved understanding of the regulation of body weight in Veteran obese patients will improve the quality of life by avoidance of serious medical complications and by suggesting novel therapeutic approaches.

The large proportion of the Veteran population that frequent the VA health care system and who suffer from obesity or have obesity-related illnesses can benefit from this research.

Obesity is associated with early mortality in the United States. It has been estimated to result in about 280,000 deaths per year in U.S. adults and the expenses related to obesity are in excess of $80 billion. Obesity is a major cause of morbidity and mortality within the VA medical system accounting for the majority of cases of diabetes mellitus, hypertension, coronary artery disease and cerebrovascular accidents.

The proposed studies will address important physiological questions regarding the mechanisms of gut peptides regulating satiety and food intake, as well as provide potentially important clinical treatment strategies. The release of GI hormones in response to meal stimuli plays an important role in the regulation of body weight homeostasis. The neural pathways interconnecting gut signaling of satiety to the brain in response to nutrient intake are regulated by neuropeptides and GI hormones.

The investigators have a long history in the study of GI hormones. In the current application, the investigators plan to elucidate the impact of a high protein diet on the profile of gut hormones released postprandially in obese subjects and the underlying changes at the neuronal (vagal afferent) level that take place in response to a high protein diet in a relevant experimental model.

Understanding the regulatory mechanisms involved in satiety will provide clues for existing and novel forms of therapies. Studies may also provide insight into underlying mechanisms responsible for weight loss induced by gastroplasty and bariatric procedure used for the treatment of obesity.

The study design is a three-group randomized, controlled study. This randomized controlled study lasting 24-30 months will assign approximately 198 volunteer subjects (ages 30, BMI 27-40 kg/m2) (66 subjects each) to the following three groups who will adhere to diets with the same number of calories:

1. Very high protein diet group based on 1.4 gram of protein per pound of lean body mass,
2. High protein diet group based on 1 gram of protein per pound of lean body mass, and
3. Standard protein diet group as control based on 0.5 gram protein per pound of lean body mass with same calories.

All participants will meet with a Registered Dietitian (who it is anticipated will join the research study team), to assist them with their diet efforts in all the arms.

In the study, the percent energy from fat will be held constant at 30% and the differences in the diets relate only to the protein and carbohydrate contents (35% protein and 35% carbohydrate, 25% protein and 45% carbohydrate, and 12.5% protein and 57.5% carbohydrate respectively).

The investigators will assess the efficacy of a high protein diet on satiety and pattern of postprandial gut hormone in obese patients. All the subjects will be followed by a dietitian and determination of circulating gut hormone and biochemical assays will be performed.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients must fulfill all of the following criteria:

* Subjects must be able to attend all 7 scheduled study visits at the West LA GI clinic at the VAGLAHS, not including the screening visit.
* Subjects must sign the VA Greater Los Angeles Healthcare System Institutional Review Board approved written informed consent prior to the initiation of any study-related activities or study specific procedures or randomization.
* Subjects must have given written authorization for the release of protected health information in compliance with Health Insurance Portability and Accountability Act (HIPAA) regulations.

After the Informed Consent process, these additional Inclusion Criteria will be applied to potential subjects:

* Age 30 years and older at screening.
* BMI of 27 to 40 kg/m2 inclusive.
* Subjects must be in good health as determined by medical history, physical examination performed by the Investigator (Study doctor) at the Screening stage, and screening clinical laboratory tests including chemistry panel and CBC.
* Must have stable smoking habits (or be non-smokers) for at least 6 months prior to screening and agree not to intend to change such habits during the course of the study.
* Subjects requiring the regular use of any prescription medication may be admitted to the study, providing the dose is stable.
* Subjects must be able to communicate and cooperate with the Principal Investigator and the staff and willing to comply with the study instructions.

Exclusion Criteria:

* Weight instability: Subjects reporting weight change of greater than 3.0 kg in the month prior to screening.
* Any subject who has been on a very low calorie diet (less than 800 kcal/day) for a period of 4 months or more in the 12 months prior to screening, or who has lost greater than 10 kg in the 6 months prior to screening.
* Any subject who has a history of diabetic gastroparesis or gastric emptying disorder as indicated in the potential subject's medical history and VA's Computer Patient Record System (CPRS).
* Use of any other investigational drug(s) within 8 weeks prior to screening.
* Subjects should not have received antibiotics within the prior 4 weeks of screening.
* Abnormal laboratory parameters:
* Serum creatinine greater than 1.6 mg/dL;
* Liver function tests, alanine transaminase (ALT), alanine transaminase (AST), Bilirubin results greater than 2.0 times the upper limit of normal;
* Triglycerides greater than 500 mg/dL;
* Total cholesterol greater than 350 mg/dL;
* Thyroid-stimulating hormone (TSH) outside of normal range disorder, as indicated in the potential subject's medical history, the VA's Computer Patient Record System (CPRS) and laboratory tests performed during the screening process.
* Subjects who drink more than 1 alcoholic beverage per day (that is: 1 beer; or 1 glass of wine; or 1 shot of liquor).
* Pregnant women or women likely to become pregnant during the course of the study may not participate in this study. Female subjects must not be able to conceive by reason of surgery, radiation, one year past the onset of menopause, or an approved method of contraception.
* No vulnerable subjects will be included in the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Pisegna, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang L, Jacobs JP, Lagishetty V, Yuan PQ, Wu SV, Million M, Reeve JR Jr, Pisegna JR, Tache Y. High-protein diet improves sensitivity to cholecystokinin and shifts the cecal microbiome without altering brain inflammation in diet-induced obesity in rats. Am J Physiol Regul Integr Comp Physiol. 2017 Oct 1;313(4):R473-R486. doi: 10.1152/ajpregu.00105.2017. Epub 2017 Jul 19. PMID 28724546
- [Background] Vu JP, Luong L, Parsons WF, Oh S, Sanford D, Gabalski A, Lighton JR, Pisegna JR, Germano PM. Long-Term Intake of a High-Protein Diet Affects Body Phenotype, Metabolism, and Plasma Hormones in Mice. J Nutr. 2017 Dec;147(12):2243-2251. doi: 10.3945/jn.117.257873. Epub 2017 Oct 25. PMID 29070713
- [Background] Stengel A, Goebel-Stengel M, Wang L, Hu E, Karasawa H, Pisegna JR, Tache Y. High-protein diet selectively reduces fat mass and improves glucose tolerance in Western-type diet-induced obese rats. Am J Physiol Regul Integr Comp Physiol. 2013 Sep 15;305(6):R582-91. doi: 10.1152/ajpregu.00598.2012. Epub 2013 Jul 24. PMID 23883680
- [Background] Vu JP, Goyal D, Luong L, Oh S, Sandhu R, Norris J, Parsons W, Pisegna JR, Germano PM. PACAP intraperitoneal treatment suppresses appetite and food intake via PAC1 receptor in mice by inhibiting ghrelin and increasing GLP-1 and leptin. Am J Physiol Gastrointest Liver Physiol. 2015 Nov 15;309(10):G816-25. doi: 10.1152/ajpgi.00190.2015. Epub 2015 Sep 3. PMID 26336928

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Diet | High Protein Diet
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Diet | High Protein Diet | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 52.69 [35 to 73] | 50.26 [32 to 71] | 51.48 [32 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 3 | 9
  White | 9 | 11 | 20
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 15 | 31
BMI [Mean (Full Range); unit: kg/m^2] | 35.49 [27 to 40] | 30.542 [27 to 40] | 33.02 [27 to 40]

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight From Baseline to 12 Months
Description: The primary objective is to compare weight loss between each of the two diets, a high-protein diet versus a standard diet.
Time Frame: The primary outcome of weight loss is measured at the Baseline at Day 1, and at the end of the 12 months study period for each subject.
Measure: Mean (Full Range); unit: lbs
Arm/Group | Standard Diet | High Protein Diet
Number analyzed (Participants) | 16 | 15
lbs | 1.09 [0 to 10] | 1.55 [0 to 10]

2. Secondary Outcome: Efficacy Variables: Nutrition Assessments (FFQ, 3DFR, and Satiety Questionnaire), Anthropometric Profiles (e.g., Waist and Hip Circumferences), Lab and Biochemical Variables (e.g., Insulin, Lipid Levels, HbA1c), Body Composition (Body Fat), Hormone Level
Description: High-protein diet promotes sensitivity to cholecystokinin and shifts the cecal microbiome without altering brain inflammation in diet-induced obesity
Time Frame: The outcome of efficacy is measured at Day 1 Baseline and at monthly visits during the 12 month study period for each subject.
Reporting Status: Not Posted

3. Secondary Outcome: Safety Variables: Incidence, Severity and Duration of Adverse Events, Vital Signs, Concomitant Medications and Physical Examination Results.
Description: as for outcome 2
Time Frame: Safety variables are measured at the time any adverse events occur, and vital signs, concomitant medications and physical examination results are measured at Baseline on Day 1 and monthly throughout the 12 month study period for each subject.
Reporting Status: Not Posted

4. Secondary Outcome: Improvement in NAFLD Fibrosis Score
Description: Patients enrolled with a history of NAFLD will be assessed for improvement in NAFLD Fibrosis scoring index and other imaging parameters if performed as standard clinical care.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Standard Diet | High Protein Diet
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT01146704/Prot_SAP_000.pdf